CLINICAL TRIAL: NCT05075967
Title: Getting to Zero Among Black Men Who Have Sex With Men (MSM) in the American South: Testing an Integrated Strategy
Brief Title: Getting to Zero Among Black MSM in the American South
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study paused due to funding
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 096
Record Dates: First submitted 2021-08-19; First posted 2021-10-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: Pre-exposure Prophylaxis (PrEP); Men who have Sex with Men (MSM); Black Men who have Sex with Men (Black MSM); HIV Incidence; Viral Suppression; Status-neutral Approach; Southern United States; Health Equity; Social Media Influencers (SMI); Intersectional Stigma Reduction; Peer Support; Black Treatment Advocates Networks (BTAN); Ending the HIV Epidemic (EHE); Black AIDS Institute (BAI); Culturally Responsive Intersectional Stigma Prevention (CRISP); Integrated Strategy; Community-randomized; Social determinants of health; Community mobilization; Community-based participatory research
MeSH Terms: conditions — HIV Infections; Homosexuality | interventions — Health Equity; Standard of Care

STUDY DESIGN:
Intervention Model Description: 16 communities will participate in the study, each made up of one or more counties selected from the southern counties and states identified in the Ending the HIV Epidemic (EHE) plan. The communities will be matched into 8 pairs based on population, HIV prevalence and viral suppression. Within each pair, one community will be randomized by public ceremony to receive the components of the integrated strategy, and the other will serve as the standard-of-care (SOC).
  A starfish sampling approach (the combination of venue-time-based and respondent-driven sampling) will be employed to recruit and enroll individual participants in both intervention and control communities for the cross-sectional assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Strategy (Experimental): Black MSM living in intervention communities will have access to the HPTN 096 integrated strategy in addition to standard HIV prevention and care services available in their communities.
  The integrated strategy includes a combination of four community-, organizational-, and interpersonal-level components designed to impact individual-level outcomes.
  Interventions: Other: Health Equity; Behavioral: Social Media Influencers; Behavioral: Intersectional Stigma Reduction; Behavioral: Peer Support
- Standard-of-care (Other): Black MSM living in standard-of-care communities will have access to standard HIV prevention and care services available in their communities.
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Other: Health Equity — This community-level structural component will use a standardized, nationally replicable community coalition model (Black Treatment Advocates Networks [BTAN]) to implement an enhanced program model geared to 1) facilitate the effects of the other HPTN 096 interventions by minimizing barriers to HIV testing, PrEP use and viral suppression through sensitizing a local network of service providers (e.g., social, legal, economic sectors) to the needs of Black MSM and maintaining an online platform for exchanging information about the local network that can be used to link Black MSM to resources and services, and 2) amplify the effects of other HPTN 096 components by increasing Black MSM's receptivity to those activities through the integration and promotion of HPTN 096 into the activities of the community coalition model.
  Arms: Integrated Strategy
Behavioral: Social Media Influencers — In this community-level component, social media influencers (SMI) will be defined for the purposes of this study as users on social media who have established credibility, trust and access to a large audience of Black MSM, and who can persuade them by virtue of their authenticity and reach. SMI will provide tailored messaging for Black MSM in intervention communities on the topics of:
  * HIV/sexually transmitted infections (STI) testing promotion
  * PrEP (and general HIV prevention) awareness and promotion
  * Definition and benefits of viral suppression.
  Messages may include direction towards health care facilities (HCFs) involved in the intersectional stigma reduction component and information about the virtual peer support platform or BTAN+ events.
  Arms: Integrated Strategy
Behavioral: Intersectional Stigma Reduction — This organizational-level component will take place in HCFs and is designed to improve cultural responsiveness in the provision of HIV prevention and health care services to Black MSM. It is expected to contribute to a reduction in HIV incidence by creating an affirming and autonomy-supportive healthcare environment that supports Black MSM engagement in HIV-related care and services and that promotes increased HIV/STI testing, PrEP uptake and viral suppression rates.
  Arms: Integrated Strategy
Behavioral: Peer Support — Peer support workers will be trained and compensated to provide emotional and practical support services. These peer support workers will have shared lived experiences with those whom they are supporting, be self-reflective of those experiences, and know when to share those experiences with others in an appropriate and supportive manner. Once trained, the peer-support workers will have demonstrated competencies in the following domains:
  * HIV, PrEP, nPEP, other HIV prevention options and ART education
  * Adherence to PrEP, ART and medical care
  * HIV/STI testing
  * New HIV diagnosis
  * Addressing intersectional stigma (anti-Black racism, sexual stigmas, HIV-related stigma)
  * Self-care
  * Information about national and local resources and assistance programs, Black MSM-centered health services, and the cost and insurance coverage of medications and medical care
  * Multicultural competency (as it relates to the HIV epidemic for Black MSM in the southern US)
  Arms: Integrated Strategy
Other: Standard-of-care — Black MSM living in standard-of-care communities will have access to standard HIV prevention and care services available in their communities.
  Arms: Standard-of-care

SUMMARY:
HPTN 096 is a community-randomized, controlled, hybrid-type III implementation effectiveness study. It is designed to evaluate an integrated strategy approach to increase the uptake and use of pre-exposure prophylaxis (PrEP) and viral suppression rates among Black MSM in the southern United States. A status-neutral approach will be taken such that Black MSM, regardless of HIV status (both those living with and without HIV), will be included in the study.

ELIGIBILITY:
The baseline and post-implementation assessment participants will be persons who:

* Self-identify as Black man (inclusive of cisgender and transgender men)
* Self-report a lifetime history of sex with other men
* Are at least 15 years of age
* Self-report current residence in the community of interest
* Are willing and able to provide informed consent
* Agree to complete a short questionnaire
* Agree to provide two blood samples (one by fingerstick and another by venipuncture).

HIV status will not be ascertained prior to participation in these assessments and eligible Black MSM may participate regardless of HIV status.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identify as a man (inclusive of cisgender and transgender men)
Enrollment: 4800 (Estimated)
Dates: Start 2022-05-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Viral suppression in Black MSM living with diagnosed HIV | Measured with data available at the end of the three year intervention
  (primary) The ratio of the number of Black MSM living with diagnosed HIV who are virally suppressed (<200 copies/mL) as measured by HIV surveillance data divided by the number of Black MSM living with diagnosed HIV as measured by HIV surveillance data
Viral suppression in Black MSM living with diagnosed HIV | Measured within six months after the end of the three year intervention
  (supportive) HIV viral load measured in the cross-sectional assessments
PrEP use by Black MSM not living with HIV | Measured within six months after the end of the three year intervention
  (primary) The presence of PrEP agents measured in a dried blood spot (DBS) collected during the cross-sectional assessments
PrEP use by Black MSM not living with HIV | Measured with data available at the end of the three year intervention
  (supportive) The ratio of the number of Black men with PrEP prescriptions (from AIDSVu) divided by the number of Black men with PrEP indications (from CDC)

SECONDARY OUTCOMES:
Self-reported HIV Testing behavior in Black MSM | Measured within six months after the end of the three year intervention
  Responses to survey questions collected during the post implementation cross-sectional assessment
Compare social support in Black MSM in the intervention to the SOC communities | Measured within six months after the end of the three year intervention
  Responses to survey questions collected during the post-implementation cross-sectional assessment
Compare intersectional stigma in Black MSM in the intervention to the SOC communities | Measured within six months after the end of the three year intervention
  Responses to survey questions collected during the post-implementation cross-sectional assessment
Compare barriers to healthcare in Black MSM in the intervention to the SOC communities | Measured within six months after the end of the three year intervention
  Responses to survey questions collected during the post-implementation cross-sectional assessment
Compare individual agency in Black MSM in the intervention to the SOC communities | Measured within six months after the end of the three year intervention
  Responses to survey questions collected during the post-implementation cross-sectional assessment
Viral suppression within 6 months of new diagnosis in Black MSM living with HIV | Measured with data available at the end of the three year intervention
  The ratio of the number of Black MSM with HIV newly diagnosed in Year 3 who have a suppressed viral load (VL) within six months of diagnosis as measured by HIV surveillance data divided by the number of Black MSM with HIV newly diagnosed in Year 3 based on HIV surveillance data
Tracking EHE implementation activities for Black MSM | Measured with data available at the end of the three year intervention
  Information about EHE implementation activities affecting Black MSM in the EHE plans of all intervention and control communities
Tracking EHE implementation activities for Black MSM | Measured with data available at the end of the three year intervention
  Information about EHE implementation activities affecting Black MSM in additional information from local health departments and EHE committees
Care quality of Black MSM needs at HCFs participating in CRISP | Measured with data available at the end of the three year intervention
  Self-reported survey data from health care workers who participate in the CRISP component
Care quality of Black MSM needs at HCFs participating in CRISP | Measured with data available at the end of the three year intervention
  Aggregated, facility-level independent ratings of HCF workers
Care quality of Black MSM needs at HCFs participating in CRISP | Measured with data available at the end of the three year intervention
  Self-reported survey data from Black MSM receiving services at HCFs participating in CRISP activities
Responsiveness to Black MSM needs at HCFs participating in CRISP | Measured with data available at the end of the three year intervention
  Self-reported survey data from health care workers who participate in the CRISP component
Responsiveness to Black MSM needs at HCFs participating in CRISP | Measured with data available at the end of the three year intervention
  Aggregated, facility-level independent ratings of HCF workers
Responsiveness to Black MSM needs at HCFs participating in CRISP | Measured with data available at the end of the three year intervention
  Self-reported survey data from Black MSM receiving services at HCFs participating in CRISP activities

CONTACTS AND LOCATIONS:
Overall Officials: LaRon Nelson, PhD, Study Chair — Yale University; Chris Beyrer, MD, Study Chair — Johns Hopkins University
Locations (1):
- FHI 360, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT05075967/Prot_000.pdf